CLINICAL TRIAL: NCT07076030
Title: Pharmacokinetics of Petrelintide Following Administration to Participants With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZP8396-24059
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 Normal Renal Function (Experimental): Each participant will receive a single subcutaneous dose of petrelintide on Day 1.
  Interventions: Drug: Petrelintide
- Group 2 Mild Renal Impairment (Experimental): Each participant will receive a single subcutaneous dose of petrelintide on Day 1.
  Interventions: Drug: Petrelintide
- Group 3 Moderate Renal Impairment (Experimental): Each participant will receive a single subcutaneous dose of petrelintide on Day 1.
  Interventions: Drug: Petrelintide
- Group 4 Severe Renal Impairment (Experimental): Each participant will receive a single subcutaneous dose of petrelintide on Day 1.
  Interventions: Drug: Petrelintide

INTERVENTIONS:
Drug: Petrelintide — Solution administered with a syringe
  Other Names: ZP8396

SUMMARY:
This clinical research study is testing the study compound petrelintide that is being developed for the weight management in people with obesity or overweight with comorbidities or related diseases.

The aim of this clinical research study is to investigate whether the effects of petrelintide will be different in people with normal kidney function compared to people with impaired kidney function.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-center, single dose, parallel-group, non-randomized study to evaluate the pharmacokinetics (PK), safety, and tolerability of petrelintide after a single dose in participants with mild, moderate, or severe renal impairment, and participants with normal renal function. Allocation of participants to the renal function groups will be based on the estimated glomerular filtration rate (eGFR).

Each participant will receive a single subcutaneous dose of petrelintide on Day 1.

Up to 24 participants with normal renal function and 24 participants with renal impairment (8 participants each in the following groups: mild, moderate, or severe renal impairment) will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65 years (both inclusive) at screening.
2. BMI (Body Mass Index): 21.0 to 40.0 kg/m2, inclusive, at screening.
3. Sex: Male and female participants.
4. Participants with mild, moderate, or severe renal impairment and participants with normal renal function.
5. For participants with renal impairment: stable renal impairment for 3 months prior to screening.
6. For participants with Type 2 diabetes mellitus and renal impairment:

   1. HbA1c (hemoglobin A1c) ≤11% at screening.
   2. On a stable diet and exercise regimen or stable metformin and/or SGLT2i (Sodium-Glucose Cotransporter 2 inhibitors) treatment for at least 3 months prior to screening.

Exclusion Criteria:

1. Exposure to amylin analogs, including petrelintide (ZP8396) within the last 3 months.
2. Clinically significant acute illness within 4 weeks prior to Day 1, as judged by the Investigator to potentially interfere with the study conduct and/or results.
3. Impaired liver function, defined as alanine aminotransferase (ALT) >1.2 times upper normal limit, or bilirubin >1.2 times upper normal limit, measured at screening.
4. Presence or history of acute or chronic pancreatitis.
5. Known clinically significant gastric emptying abnormality (for example, severe gastroparesis, gastric outlet obstruction, gastric bypass operations, or sleeve gastrectomies) or chronic treatment that affects gastrointestinal motility.
6. Any disorder, unwillingness, or inability, not covered by any of the other exclusions criteria, which in the Investigator´s opinion, might jeopardize the participant´s safety or compliance with the protocol.
7. Participants with Type 1 diabetes mellitus as declared by the participant.
8. A history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
9. Presence or history of clinically significant arrhythmias or clinically significant conduction disorders.
10. A marked baseline prolongation of QT/QTc (e.g. repeated demonstration of a QTc interval >450 ms.
11. Smoking of more than 10 cigarettes (or equivalent nicotine consumption) per day.

    Tobacco that contains menthol must not be consumed within 7 days prior to study drug administration.
12. Presence or history of following cardiovascular diseases:

    1. Decompensated heart failure (New York Heart Association (NYHA) class III and IV).
    2. Unstable angina pectoris.
    3. Myocardial infarction within the last 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
AUCo-inf of petrelintide | From administration (Day 1) to Last visit (Day 43)
  AUCo-inf: Area Under the Curve from time 0 to infinity

SECONDARY OUTCOMES:
Maximum observed plasma concentration | From administration (Day 1) to Last visit (Day 43)
Time to attain maximum observed plasma concentration | From administration (Day 1) to Last visit (Day 43)
Area under the plasma concentration-time curve from time 0 to infinity | From administration (Day 1) to Last visit (Day 43)
Area under the concentration versus time curve from time zero to last measurable concentration | From administration (Day 1) to Last visit (Day 43)
Terminal elimination half-life | From administration (Day 1) to Last visit (Day 43)
Apparent clearance | From administration (Day 1) to Last visit (Day 43)
Apparent volume of distribution at terminal phase | From administration (Day 1) to Last visit (Day 43)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Kegel-Hübner, Dr.med., Principal Investigator — Charité Research Organisation GmbH
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No